CLINICAL TRIAL: NCT00142376
Title: Short Term Outcomes of Children With Acute Respiratory Distress Syndrome
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Other Study IDs: 0409HSE222
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2005-09-02 (Estimated); Status verified 2004-09

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
The study is a chart review of all children admitted over a two year period with the diagnosis of acute respiratory distress syndrome. Short term outcomes, such as mortality, length of ventilation and length of stay, will be reviewed. Factors that impact these outcomes will also be reviewed.

DETAILED DESCRIPTION:
We would like to conduct a chart review of all patients with pediatric ARDS hospitalized in the PICU at Columbus Children's Hospital in the last two years. Patients would be included for review if they met the clinical criteria for ARDS. These criteria are: rapidly progressive respiratory failure, severe hypoxemia (PaO2/FiO2 < 200), and evidence of bilateral pulmonary infiltrate on chest radiography. We estimate 40-50 patients will meet criteria.

Once criteria are met, patient charts will be pulled or reviewed electronically. We will then compose a database that includes no patient identifiers but contains information regarding the cause, length, and outcome of the ARDS admission and PICU stay. Factors such as nutritional status, antibiotic and muscle relaxant use, and type of ventilation used will be examined. Other care-related variables will be included if they are felt to impact outcome during the review process. The database will then be analyzed and information regarding pediatric ARDS outcomes in our institution will be published.

We anticipate that examining the factors that impact short term outcomes in pediatric ARDS will lead to research possibilities regarding ways to improve both short and long term outcomes in children with this illness. We propose that reviewing the disease entity as a whole will lead to improvements in caring for children with the disease, and eventually bring about a decline in mortality rates.

ELIGIBILITY:
Inclusion Criteria:

* Rapidly progressive respiratory failure,
* Severe hypoxemia (PaO2/FiO2 < 200),
* Evidence of bilateral pulmonary infiltrate on chest radiography
* 0-18 years of age

Exclusion Criteria:

* Heart failure
* Cardiac shunt present

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2004-09; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Onsy Ayad, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Columbus Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Bernard GR, Artigas A, Brigham KL, Carlet J, Falke K, Hudson L, Lamy M, Legall JR, Morris A, Spragg R. The American-European Consensus Conference on ARDS. Definitions, mechanisms, relevant outcomes, and clinical trial coordination. Am J Respir Crit Care Med. 1994 Mar;149(3 Pt 1):818-24. doi: 10.1164/ajrccm.149.3.7509706.
- [Background] Davis SL, Furman DP, Costarino AT Jr. Adult respiratory distress syndrome in children: associated disease, clinical course, and predictors of death. J Pediatr. 1993 Jul;123(1):35-45. doi: 10.1016/s0022-3476(05)81534-3. PMID 8320623
- [Background] Timmons OD, Havens PL, Fackler JC. Predicting death in pediatric patients with acute respiratory failure. Pediatric Critical Care Study Group. Extracorporeal Life Support Organization. Chest. 1995 Sep;108(3):789-97. doi: 10.1378/chest.108.3.789. PMID 7656635
- [Background] Katz R. Adult respiratory distress syndrome in children. Clin Chest Med. 1987 Dec;8(4):635-9. PMID 3322648
- [Background] Timmons OD, Dean JM, Vernon DD. Mortality rates and prognostic variables in children with adult respiratory distress syndrome. J Pediatr. 1991 Dec;119(6):896-9. doi: 10.1016/s0022-3476(05)83039-2. PMID 1960603
- [Background] Milberg JA, Davis DR, Steinberg KP, Hudson LD. Improved survival of patients with acute respiratory distress syndrome (ARDS): 1983-1993. JAMA. 1995 Jan 25;273(4):306-9. PMID 7815658
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162